CLINICAL TRIAL: NCT05018611
Title: Digital, Limited Interaction Efficacy Trial of LifeSkills Mobile to Reduce HIV Incidence in Young Transgender Women
Brief Title: Digital Limited Interaction Efficacy Trial of LifeSkills Mobile to Reduce HIV Incidence in YTW
Acronym: LifeSkills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, ScD, MPH, MA, Professor of Epidemiology, UCLA Fielding School of Public Health, and Psychiatry & Biobehavioral Sciences, UCLA David Geffen School of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 U01 A1156875
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: HIV Prevention
Keywords: Transgender women (TGW); PrEP; mHealth; HIV Prevention; Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LifeSkills Mobile (Experimental): Access to LifeSkills Mobile app. Participants will complete 4 modules with 20 activities across 6 months. Participants can log in at their convenience but will not be able to access the next module until the previous module is completed.
  Interventions: Behavioral: LifeSkills Mobile
- Standard of Care (No Intervention): HIV home testing every 6 months, information regarding sexual and other behaviors that potentiate one's risk for HIV infection, receipt of a fact sheet about PrEP and PEP and referrals to the local PrEP clinics, and sexually transmitted infection testing via an on-line location findings app.

INTERVENTIONS:
Behavioral: LifeSkills Mobile — A mobile app designed to facilitate the broad reach and impact of the LifeSkills intervention to reduce sexual risk behavior which drives HIV infection. The LifeSkills intervention addresses the specific structural, developmental, and interpersonal challenges to HIV prevention among YTW ages 16-29, with prior evidence of the efficacy to reduce sexual risk.
  Arms: LifeSkills Mobile

SUMMARY:
The LifeSkills Mobile app will be evaluated in a randomized controlled trial (RCT) among 5,000 young transgender women (YTW), ages 16-29 in the United States (U.S.). Study findings will demonstrate if the intervention will reduce HIV incidence.

DETAILED DESCRIPTION:
LifeSkills Mobile is an mHealth intervention to promote biobehavioral HIV prevention strategies based on empowerment theory and was developed using a community-based participatory research approach. An RCT assesses the efficacy of the LifeSkills Mobile intervention in comparison to a standard of care (SOC) condition among 5,000 YTW recruited online. At baseline and every 6 months through 12-48 months (depending on when the participant enrolled), enrolled participants will complete an online survey sent via a link to their mobile phone and will be mailed an OraQuick In-Home HIV Test kit. We will also estimate the total and incremental costs of the LifeSkills Mobile intervention relative to SOC, from healthcare sector and societal perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as transgender, woman, and/or along the feminine spectrum with a male assigned sex at birth
* Ages 16-29
* HIV uninfected at enrollment visit, verified via HIV home test kit
* Self-reported lifetime history of condomless sex or recent history of sex (anal or vaginal in the past 12 months)
* Able to speak/understand English
* Owns a smartphone or home computer or willing to use one in the study
* Willing and able to provide informed consent/assent

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at time of enrollment
* Discovery of active suicidal ideation or major mental illness (e.g. untreated psychosis or mania) at the time of the interview (these patients will be referred immediately for treatment, but may join the study when this is resolved)
* A positive Home HIV test kit result at baseline; these individuals will be immediately linked to HIV clinical care in their local areas.

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identified as transgender, woman, and/or along the feminine spectrum
Enrollment: 5100 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
HIV incidence | 12-48 months post-baseline (depending on when participants enroll in the study)
  Participants will be mailed and take an OraQuick In-Home HIV Test. Reactive HIV screening tests will be confirmed via dried blood spot (DBS; detectable antibodies). The main analysis will assess whether there are differences in survival (or cumulative incidence of HIV) among those randomized to LifeSkills Mobile versus those randomized to SOC.

SECONDARY OUTCOMES:
Changes in sexual risk behavior at 6 months based on self-report | 6 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 12 months based on self-report | 12 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 18 months based on self-report | 18 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 24 months based on self-report | 24 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 30 months based on self-report | 30 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 36 months based on self-report | 36 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 42 months based on self-report | 42 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Changes in sexual risk behavior at 48 months based on self-report | 48 months post-baseline
  Self-reported total condomless anal or vaginal sex acts in the prior 30 days without protection via PrEP
Comparison of costs between LifeSkills Mobile intervention vs SOC | End of study
  Total and incremental costs of the LifeSkills Mobile intervention relative to SOC, from healthcare sector and societal perspectives
PrEP outcomes (linkage, initiation, retention) | 12-48 months post-baseline (depending on when participants enroll in the study)
  PrEP care linkage defined as attending at least one PrEP-related care visit to assess medical eligibility for PrEP initiation in the prior 6 months, per self-report PrEP initiation defined as starting PrEP medication in the prior 6-month period by self-report PrEP retention defined as: at least one PrEP care visit in a 6-month period PrEP visit constancy defined as at least one visit every six months over a 12-month period per self-report

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Belzer, MD, Principal Investigator — Children's Hospital Los Angeles; Matthew J Mimiaga, ScD, MD, Principal Investigator — University of California, Los Angeles; Lisa Kuhns, PhD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhns LM, Garofalo R, Belzer M, McAvoy-Banerjea J, Holzman J, Kwak E, Johnson AK, Biello K, Schnall R, Hidalgo MA, Reisner SL, Mimiaga MJ. Digital limited interaction efficacy trial of LifeSkills Mobile to reduce HIV incidence in young transgender women: study protocol. Trials. 2025 Dec 17. doi: 10.1186/s13063-025-09353-0. Online ahead of print. PMID 41402905